CLINICAL TRIAL: NCT05824221
Title: Effect of rTMS on BDNF and proBDNF Levels: a Sham-controlled Study in Subjects With Cocaine Use Disorder
Brief Title: Effect of rTMS on Neurotrophines Levels in CUD
Acronym: BDNFcoca
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Mauro Pettorruso, Principal Investigator, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: brainbdnf
Record Dates: First submitted 2023-04-05; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cocaine Use; Cocaine Dependence; Cocaine Abuse; Neurotropism
Keywords: rTMS; BDNF; proBDNF; Cocaine Use Disorder
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Intervention Model Description: randomized, sham-controlled with a 1:1 allocation into 2 parallel arms. A third arm constituted by healthy patients.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With regard to the treatment, to ensure that both participants and investigators are blind to the condition (active or sham), the selection of the operation mode (15 Hz, sham) will be pre-programmed by member of the that will not be involved in data collection and analysis. Study personnel will not know which mode is being activated. Sham stimulation will use the same coil placement as that used for active stimulation. Outcomes Assessors will not be present during the rTMS sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active rTMS (15 Hz) (Experimental): Active stimulation of LDLPFC (15 Hz; 100% of RMT; 40 trains with 60 stimuli per train; inter-train interval of 15 second, total duration 13 minutes). Each session will be repeated twice/daily for 10 consecutive days for 2 weeks, during the continued treatment phase. Device: MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): A pre-programmed software set sham stimulation by a staff member that will not be involved in data collection and analysis. The sham condition will match the number of pulses delivered during the 15Hz session and will use the same coil placement but the intensity of stimulation will be set a 3% of the RMT so to ensure that the participant will feel similar scalp sensations experienced by participants receiving active rTMS, but brain tissue will not be stimulated. Device: MagPro R30 with the Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Interventions: Device: rTMS
- Healthy Control (No Intervention): Subject without diagnosis of Cocaine Use Disorder or other major psychiatric disorder.

INTERVENTIONS:
Device: rTMS — Non invasive brain stimulation in Cocaine Use Disorder
  Arms: Active rTMS (15 Hz); Sham rTMS

SUMMARY:
Brief Summary:

Background: Cocaine use disorders (CUD) is a multifactoral disease, involving several brain areas. One of the most investigated is the Dorsolateral Prefrontal Cortex (DLPFC) involved in impulsiveness control. Effective treatments for CUD are still needed and repetitive Transcranial Magnetic Stimulation (rTMS) is widely studied for its potential in reducing cocaine craving and consumption.

Objectives: The main outcome is to test if rTMS can be related to neuroplasticity and neurotrophism through changes in Brain-Derived Neurotrophic Factor (BDNF) and its precursor (pro-BDNF) levels.

Eligibility: Healthy, right-handed adults ages 18-65 who do have cocaine use disorder (moderate to severe).

Design: This is a randomized, sham-controlled study. The study includes a rTMS continued treatment phase compared to healthy control (HC) evaluation.

Prior to participating, participants will be screened with:

* Medical history
* Anamnestic sheet
* Physical exam
* Urine tests After being enrolled, participants and HC will undergo venous blood sample (BDNF and proBDNF levels).

During the continued rTMS phase, participants with cocaine use disorder will be randomized to receive real or sham rTMS; a former arm is also provided and is made up of HC. RTMS will be delivered in 10 days, over 2 weeks (5 days/week). After the last rTMS session a blood sample for neurotrophines levels will be collected.

Treatment includes:

* rTMS: A coil is placed on the head. At each session, participants will receive two rTMS sessions, with a 50 mins interval. At the beginning of each rTMS session, they view cocaine-related images for few minutes (cue-induced stimuli).
* BDNF/proBDNF levels: A venous blood sample will be collected before the first stimulation and after the last stimulation of the intensive-stimulation period (first two weeks), this sample will be also collected from HC. The blood sample will be centrifuged within 20 minutes of sampling at 1000 × g for 15 minutes. Then, the serum will be aliquoted and stored at -80 ° C until analysis.
* Urine toxicological screen

DETAILED DESCRIPTION:
RTMS has been shown to reduce craving in CUD. The purpose of this study is to assess the effects of rTMS at 15 Hz frequency on neurotrophines serum levels . For this purpose, the investigators will recruit cocaine user. After screening and informed consent, participants will undergo active or sham rTMS for two consecutive weeks (twice a day) during the continued treatment phase; a third arm of HC will receive no treatment. A venous blood sample will be collected before the first stimulation and after the last stimulation of the first two weeks treatment.

Procedure: The project consists of: Screening Visit (baseline) and the continued treatment phase, In the screening visit, a clinical interview to assess the eligibility of participant (following the inclusion and exclusion criteria) will be performed. All participants will be randomly assigned to one of the two treatment arms with rTMS (15Hz, 15Hz-Sham). Participants will receive 2 sessions of rTMS (active or sham), twice per day for 10 consecutive days, for a total of 20 rTMS sessions. A venous blood sample will be collected before the first stimulation and after the last stimulation of the continued treatment phase to asses the BDNF and pro-BDNF level.

ELIGIBILITY:
Inclusion Criteria (for CUD patient):

1. Current diagnosis of cocaine use disorder (from moderate to severe), based on the Diagnostic and Statistical Manual of Mental Disorder - Fifth Edition (DSM-5);
2. Abstinence from cocaine for at least 48 hrs.

Exclusion Criteria (for CUD patient):

1. Current DSM-5 diagnosis of substance and/or alcohol use disorders other than nicotine;
2. Current DSM-5 diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder;
3. Use in the past 4 weeks of any medication with known pro-convulsant action; or current regular use of any psychotropic medications (benzodiazepines, antipsychotic medications, tricyclic antidepressants, anti-epileptics, mood stabilizers);
4. Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;

Inclusion Criteria (for HC):

1. 18-65 years

Exclusion Criteria (for CUD patient):

1. Current DSM-5 diagnosis of substance use disorders other than nicotine;
2. Current DSM-5 diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in BDNF level (biological marker) | Baseline, two weeks
  BDNF levels will be evaluated by collecting a venous blood sample. BDNF is a member of the nerve growth factor (NGF) family of neurotrophic growth factors. The increase in serum levels of BDNF seems to reflect the neuroplasticity of the CUD brain. BDNF measurements will be calculated in pg/ml
Change in proBDNF level (biological marker) | Baseline, two weeks
  Pro-BDNF is the precursor of BDNF and it acts as a repository of mature BDNF and acts itself by inducing neuronal thinning. Pro-BDNF levels will be evaluated by collecting a venous blood sample. Pro-BDNF measurements will be calculated in ng/ml.
Change in pro-BDNF/BDNF ratio (biological marker) | Baseline, two weeks
  Pro-BDNF/BDNF ratio, seems to be a more specific measurement of the early changes in the metabolism of BDNF. Its level seems to correlate to more or less a neurotrophic and neuroprotective action of BDNF. As a ratio it has not a unit measure.

CONTACTS AND LOCATIONS:
Locations (1):
- ITAB, Chieti, Italy

IPD SHARING:
Plan to Share IPD: No